CLINICAL TRIAL: NCT02950805
Title: A Phase 1b Randomized Blinded Placebo-Controlled, Cross-Over Study to Assess the Effect of AZD5634 on Mucociliary Clearance as Well as Safety, Tolerability, and Pharmacokinetic Parameters Following Single Inhaled Dose Administration to Patients With Cystic Fibrosis.
Brief Title: A Study to Assess the Effect of AZD5634 on Mucociliary Clearance, Safety, Tolerability and Pharmacokinetic Parameters in Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6600C00002
Record Dates: First submitted 2016-08-23; First posted 2016-11-01 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Pulmonary/Respiratory Diseases
Keywords: AZD5634; Mucociliary Clearance; Safety; Tolerability; Pharmacokinetic; Cystic Fibrosis; Cross-Over Study
MeSH Terms: conditions — Respiratory Tract Diseases; Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo + AZD5634 (Experimental): Subjects were administered single dose of placebo in period 1 and AZD5634 in period 2.
  Interventions: Drug: Placebo; Drug: AZD5634
- AZD5634 + Placebo (Experimental): Subjects were administered single dose of AZD5634 in period 1 and placebo in period 2.
  Interventions: Drug: Placebo; Drug: AZD5634

INTERVENTIONS:
Drug: Placebo — Subjects will receive a placebo in either period 1 or period 2 by inhalation.
Drug: AZD5634 — Subjects will receive a single tentative dose of 625 μg of AZD5634 in either period 1 or period 2 by inhalation.

SUMMARY:
This study will assess the effect of inhaled AZD5634 on Mucociliary clearance (MCC) in patients with Cystic fibrosis (CF) after single-dose administration.

DETAILED DESCRIPTION:
The primary pharmacodynamic endpoint will be the average whole lung particle clearance between 0 and 60 minutes after administration of aerosolized radiolabelled particles (colloids) at Visits 2 and 3 (%MCC 0-60, whole).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated written informed consent prior to any study-specific procedures.
2. Male or female patients aged 18-60 years old inclusive.
3. Diagnosed of CF at Screening as evidenced in medical records by one of the following criteria:

   1. sweat chloride ≥ 60 mmol/L
   2. presence of 2 mutations in the Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) gene.
4. Chronic sinopulmonary disease or pancreatic insufficiency.
5. FEV1measurement at Screening ≥ 40% of the predicted normal value of age, height, gender, and race.
6. Stable CF regimen for at least 2 months before Screening.
7. Body mass index (BMI) between 15-30 kg/m2 inclusive.
8. Female patients are not pregnant and do not plan to become pregnant during the study, are not lactating, or are of non-childbearing potential. Females of childbearing potential must provide a negative serum pregnancy test and have a date of last menstruation consistent with non-pregnancy, negative urine pregnancy tests at each visit, and must be using at least one highly effective method of contraception.
9. Ability of the patient to correctly perform the inhalation procedure after training during the Screening Visit.

Exclusion Criteria:

1. Had a pulmonary exacerbation requiring change in antibiotics and/or hospitalization within 28 days before the first dose of Investigational product.
2. History of lung transplant or any other transplantation.
3. Currently being treated with ivacaftor monotherapy at Screening or received ivacaftor monotherapy within 30 days before Screening.
4. History of severe allergy/hypersensitivity or ongoing clinically significant allergy/hypersensitivity, as judged by the Investigator, to drugs in a similar class to AZD5634.
5. History or presence of hepatic cirrhosis.
6. Creatinine clearance <60 mL/min/m2 using the Cockroft-Gault Equation.
7. Liver function test results >2x upper limit of normal (aspartate aminotransferase [AST], alanine aminotransferase [ALT], gamma-glutamyl transpeptidase [GGT], or bilirubin)
8. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study, or influence the results or the patient's ability to participate in the study.
9. Received treatment with the following medications within the 3 weeks before Screening: strong or moderate Cytochrome P450 (CYP) 3A inhibitors, as classified by the Food and Drug Administration (FDA).
10. Likely to require treatment during the study with drugs not permitted by the study protocol.
11. Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results.
12. Serum potassium levels are outside the normal range (3.5-5.1 mmol/L).
13. Serum sodium levels <135 mmol/L.
14. Abnormal vital signs, after 5 minutes rest, at Screening or Visit 2 (seated or supine; position should be consistent for a given patient at both visits), defined as any of the following:

    * Systolic blood pressure (B.P) < 90 or ≥ 150 mmHg
    * Diastolic B.P < 45 or ≥ 90 mmHg
    * Pulse rate < 45 or >110 beats/minute
15. Any clinically significant abnormalities in rhythm, conduction, or morphology of the resting ECG and any clinically significant abnormalities in the 12-lead ECG, as considered by the Investigator, that may interfere with the interpretation of corrected ECG interval measured from the onset of the QRS complex to the offset of the T wave (QTc) interval changes.
16. QTc prolongation defined as QT interval corrected for heart rate using Fridericia's formula (QTcF) >450 ms.
17. ECG interval measured from the onset of the P wave to the onset of the QRS complex (PR/PQ) interval prolongation (>240 ms), intermittent second or third degree atrioventricular (AV) block, or AV dissociation.
18. Persistent or intermittent complete bundle branch block (BBB) with ECG interval measured from the onset of the QRS complex to the J point (QRS) >120 ms or evidence of pre-excitation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-04-12 (Actual)

PRIMARY OUTCOMES:
Percentage of average whole lung particle clearance between 0 and 60 minutes after administration of aerosolized radiolabelled particles | 0 to 60 minutes
  Assessment of the average whole lung clearance between 0 and 60 minutes after administration of single inhaled dose of aerosolized radiolabelled particles (colloids) of AZD5634, (%MCC 0--60, whole) in subjects with cystic fibrosis (CF).

SECONDARY OUTCOMES:
Percentage of average central clearance between 0 and 60 minutes after administration of aerosolized radiolabelled particles | 0 to 60 minutes
  Assessment and comparison of the average central clearance between 0 and 60 minutes after administration of single inhaled dose of aerosolized radiolabelled particles (colloids) of AZD5634, in subjects with CF.
Percentage of average peripheral clearance between 0 and 60 minutes after administration of aerosolized radiolabelled particles | 0 to 60 minutes
  Assessment and comparison of the average peripheral clearance between 0 and 60 minutes after administration of single inhaled dose of aerosolized radiolabelled particles (colloids) of AZD5634 in subjects with CF.
Percentage of average tracheobronchial clearance between 0 and 60 minutes after administration of aerosolized radiolabelled particles | 0 to 60 minutes
  Assessment and comparison of the average tracheobronchial clearance between 0 and 60 minutes after administration of single inhaled dose of aerosolized radiolabelled particles (colloids) of AZD5634 in subjects with CF.
Percentage of particle clearance at 6-hour | 6 hours
  Assessment and comparison the 6-hour clearance after administration of aerosolized radiolabelled particles (colloids) of AZD5634 in subjects with CF.
Percentage of average whole lung cough clearance between 60 minutes and 90 minutes after administration of aerosolized radiolabelled particles | 60 minutes to 90 minutes
  Assessment of the average whole lung cough clearance between 60 minutes and 90 minutes after administration of single inhaled dose of aerosolized radiolabelled particles (colloids) of AZD5634 in subjects with CF.
Percentage of average central cough clearance between 60 minutes and 90 minutes after administration of aerosolized radiolabelled particles | 60 minutes to 90 minutes
  Assessment and comparison of the average central cough clearance between 60 minutes and 90 minutes after administration of single inhaled dose of aerosolized radiolabelled particles (colloids) of AZD5634 in subjects with CF.
Percentage of average peripheral cough clearance between 60 minutes and 90 minutes after administration of aerosolized radiolabelled particles | 60 minutes to 90 minutes
  Assessment and comparison of the average peripheral cough clearance between 60 minutes and 90 minutes after administration of single inhaled dose of aerosolized radiolabelled particles (colloids) of AZD5634 in subjects with CF.
Percentage of average tracheobronchial cough clearance between 60 minutes and 90 minutes after administration of aerosolized radiolabelled particles | 60 minutes to 90 minutes
  Assessment and comparison of the average tracheobronchial cough clearance between 60 minutes and 90 minutes after administration of single inhaled dose of aerosolized radiolabelled particles (colloids) of AZD5634 in subjects with CF.
Maximum observed plasma concentration (Cmax) | Pre-dose and up to 6 hours post-dose
  Assessment of Cmax in subjects with CF after the administration of single inhaled dose of AZD5634.
Area under the concentration-time curve from time zero extrapolated to infinity (AUC) | Pre-dose and up to 6 hours post-dose
  Assessment of AUC in subjects with CF after the administration of single inhaled dose of AZD5634.
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC 0-last) | Pre-dose and up to 6 hours post-dose
  Assessment of AUC 0-last in subjects with CF after the administration of single inhaled dose of AZD5634.
Area under the plasma concentration-time curve from time zero to 6 hours post-dose (AUC 0-6) | Pre-dose and up to 6 hours post-dose
  Assessment of AUC 0-6 in subjects with CF after the administration of single inhaled dose of AZD5634.
Observed last quantifiable concentration (C last) | Pre-dose and up to 6 hours post-dose
  Assessment of C last in subjects with CF after the administration of single inhaled dose of AZD5634.
Time of last quantifiable concentration (t last) | Pre-dose and up to 6 hours post-dose
  Assessment of t last in subjects with CF after the administration of single inhaled dose of AZD5634.
Time to reach maximum plasma concentration (t max) | Pre-dose and up to 6 hours post-dose
  Assessment of t max in subjects with CF after the administration of single inhaled dose of AZD5634.
Terminal elimination rate constant (λz) | Pre-dose and up to 6 hours post-dose
  Assessment of λz in subjects with CF after the administration of single inhaled dose of AZD5634.
Terminal elimination half-life (t1/2,λz) | Pre-dose and up to 6 hours post-dose
  Assessment of t1/2,λz in subjects with CF after the administration of single inhaled dose of AZD5634.
Apparent clearance (CL/F) | Pre-dose and up to 6 hours post-dose
  Assessment of CL/F in subjects with CF after the administration of single inhaled dose of AZD5634.
Apparent volume of distribution at terminal phase (Vz/F) | Pre-dose and up to 6 hours post-dose
  Assessment of Vz/F in subjects with CF after the administration of single inhaled dose of AZD5634.
Cumulative amount of AZD5634 excreted in urine from time zero to 6 hours (Ae 0-6) | Pre-dose and up to 6 hours post-dose
  Assessment of Ae 0-6 in subjects with CF after the administration of single inhaled dose of AZD5634.
Cumulative percentage of dose excreted unchanged in urine from time zero to 6 hours (fe(0-6)%) | Pre-dose and up to 6 hours post-dose
  Assessment of fe(0-6)% in subjects with CF after the administration of single inhaled dose of AZD5634.
Renal clearance, estimated by dividing Ae(0-t) (CLR) | Pre-dose and up to 6 hours post-dose
  Assessment of CLR in subjects with CF after the administration of single inhaled dose of AZD5634.
  CLR is defined as renal clearance, estimated by dividing Ae(0-t) cumulative amount of AZD5634 excreted in urine from time zero up to time t) by AUC 0-t (area under the plasma concentration-time curve from time zero to time t), where t represents a matching time point for plasma and urine sampling.
Safety of subjects by evaluating the incidence of adverse events (AEs) | From screening (≤28 days) up to 14-21 days post dosing
  Assessment of the safety in terms of the incidences of the AEs after the administration of single inhaled dose of AZD5634 in subjects with CF.
Safety of subjects by evaluating the systolic and diastolic blood pressure | From screening (≤28 days) up to 14-21 days post dosing
  Assessment of the safety in terms of systolic and diastolic blood pressure after the administration of single inhaled dose of AZD5634 in subjects with CF.
Safety of subjects by evaluating the pulse rate. | From screening (≤28 days) up to 14-21 days post dosing
  Assessment of the safety in terms of pulse rate after the administration of single inhaled dose of AZD5634 in subjects with CF.
Safety of subjects by evaluating spirometry results | From screening (≤28 days) up to 14-21 days post dosing
  Assessment of the safety by evaluating the spirometry results after administration of the of single inhaled dose of AZD5634 in subjects with CF.
Safety of subjects by evaluating the ECG results | Pre-dose and up to 6 hours post-dose
  Assessment of the safety by evaluating the ECG results after administration of the of single inhaled dose of AZD5634 in subjects with CF.
Safety of subjects by the physical examination | From screening (≤28 days) up to 14-21 days post dosing
  Assessment of the safety by physical examination after administration of the of single inhaled dose of AZD5634 in subjects with CF.
Safety of subjects by evaluating the respiratory rate. | From screening (≤28 days) up to 14-21 days post dosing
  Assessment of the safety in terms of respiratory rate after the administration of single inhaled dose of AZD5634 in subjects with CF.
Safety of subjects by evaluating fractional excretion of potassium (FEK) | Pre-dose and at 0-6 hours post-dose
  Assessment of FEK after the administration of single inhaled dose of AZD5634 in subjects with CF.
Safety of subjects by evaluating urine sodium/potassium (Na/K) ratio | Pre-dose and at 0-6 hours post-dose
  Assessment of ratio of Na/K after the administration of single inhaled dose of AZD5634 in subjects with CF.
Safety of subjects by evaluating the pulse oximetry | From screening (≤28 days) up to 14-21 days post dosing
  Assessment of the safety in terms of pulse rate after the administration of single inhaled dose of AZD5634 in subjects with CF.
Safety of subjects by evaluating the clinical laboratory test results for biochemistry | From screening (≤28 days) until 14-21 days post dosing
  Assessment of the clinical laboratory test results in terms of biochemistry after the administration of single inhaled dose of AZD5634 in subjects with CF.
Safety of subjects by evaluating the clinical laboratory test results for urinalysis | From screening (≤28 days) until 14-21 days post dosing
  Assessment of the clinical laboratory test results in terms of urinalysis after the administration of single inhaled dose of AZD5634 in subjects with CF.
Safety of subjects by evaluating the clinical laboratory test results for hematology | From screening (≤28 days) until 14-21 days post dosing
  Assessment of the clinical laboratory test results in terms of hematology after the administration of single inhaled dose of AZD5634 in subjects with CF.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Research Site, Birmingham, Alabama
  - Research Site, Baltimore, Maryland
  - Research Site, Chapel Hill, North Carolina

REFERENCES:
- [Derived] Kristensson C, Astrand A, Donaldson S, Goldwater R, Abdulai R, Patel N, Gardiner P, Tehler U, Mercier AK, Olsson M, Ersdal E, Maenpaa J, Bramer T, Malmgren A, Bennett W, Keen C. AZD5634, an inhaled ENaC inhibitor, in healthy subjects and patients with cystic fibrosis. J Cyst Fibros. 2022 Jul;21(4):684-690. doi: 10.1016/j.jcf.2022.02.010. Epub 2022 Feb 26. PMID 35227647